CLINICAL TRIAL: NCT01584297
Title: Open Phase II Study of Ketoconazole as Inhibitor of the Enzyme CYP17 in Locally Advanced or Disseminated Granulosa Cell Tumour of Ovary. GreKo Study.
Brief Title: Ketoconazole as Inhibitor of the Enzyme CYP17 in Locally Advanced or Disseminated Granulosa Cell Tumour of Ovary
Acronym: GreKo
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient recruitment rate
Sponsor: Grupo Español de Tumores Huérfanos e Infrecuentes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GETHI 2011-03; 2012-001948-21 (EudraCT Number)
Record Dates: First submitted 2012-04-22; First posted 2012-04-24 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Granulosa Cell Tumour of the Ovary
Keywords: Granulosa Cell Tumour
MeSH Terms: conditions — Granulosa Cell Tumor | interventions — Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ketoconazole (Experimental): Patients will receive ketoconazole, 400 mg three times a day. Study treatment period will be during 6 months or up to progression disease, unacceptable toxicity, death or withdraw from the study for any reason.
  Interventions: Drug: Ketoconazole

INTERVENTIONS:
Drug: Ketoconazole — Patients will receive ketoconazole, 400 mg three times a day. Study treatment period will be during 6 months or up to progression disease, unacceptable toxicity, death or withdraw from the study for any reason.
  Other Names: Fungarest

SUMMARY:
Our proposal is to conduct an open phase II clinical trial that allows us to explore the activity of ketoconazole, an inhibitor of the enzyme CYP17, in ovarian granulosa tumors similar to what has been done in prostate cancer. The rational is based on dysregulation that FOXL2 mutations present in almost all granulosa tumors result in the expression of CYP17 that appears to be key in the development and progression of the disease.

This work would represent the first attempt to address the treatment of ovarian granulosa cancer with a molecular solid rational, drawing on the recent identification of the mutation "leader" of this tumor. If succeed provide a widely available therapeutic alternative compared with current cancer therapies, with low toxicity. In addition it would open a new line of research with CYP17 enzyme inhibitors that could alter the course and outcome, usually fatal, in advanced stages of disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients obtained their written informed consent.
* Women ≥18 years old.
* ECOG ≤ 1.
* Histologically confirmed carcinoma of granulosa cell in ovary.
* Availability of sufficient biopsy material to confirm the diagnosis by a centralized pathologist and determination of the FOXL2 402C mutation → G (C134W).
* Metastatic or unresectable disease.
* Imaging measurable disease.
* Life expectancy ≥ 12 weeks.
* Patients with adequate hepatic function, defined by:
* Serum values of AST and ALT ≤ 3 x UNL (except in the presence of metastases then allowed values ≤ 5 x UNL)
* Total bilirubin ≤ 1.5 x UNL
* Patients with adequate bone marrow function, defined by:
* Absolute neutrophil count ≥ 1.5 x 10*9 / L
* Platelets ≥ 100 x 10*9 / L
* Hb > 9 g / dL
* Patients with adequate renal function: serum creatinine ≤ 1.5 x UNL.
* Absence of any impediment to comply with the study protocol.
* Women of childbearing potential, sexually active, not under hysterectomy or bilateral adnexectomy, should follow the following guidelines on contraception:
* Negative serum or urine pregnancy test within 72 hours before the start of treatment.
* Use of a medically accepted contraceptive method during: the 2 months prior to study treatment, during the study and 3 months after the last dose of study treatment.

Exclusion Criteria:

* Patients with another primary tumor 2 years before starting the study drug, with the exception of cervical carcinoma in situ or adequately treated or removed completely or basalioma or superficial bladder carcinoma.
* Patients received radical radiotherapy ≤ 4 weeks before starting the study treatment or who have not recovered from the toxicities of radiotherapy. Palliative radiotherapy of painful bone lesions is allowed up to 14 days before the start of study treatment.
* Patients with heart failure or clinically significant heart disease, including any of the following:
* History or presence of uncontrolled severe ventricular arrhythmia.
* Clinically significant bradycardia at rest.
* LVEF <45% assessed by 2-D echocardiogram (ECHO) or MUGA.
* Any of the following diseases within 6 months prior to the start of study drug: Myocardial infarction (MI), severe or unstable angina, coronary revascularization, congestive heart failure (CHF), stroke (CVA), transient ischemic attack (TIA).
* Patients with gastrointestinal function failure or gastric disease that significantly alter the ketoconazole absorption, for example, severe ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption, extensive resection (> 1m) of the small intestine or inability to swallow oral medication. The partial or total gastrectomy is not an exclusion criteria.
* Diagnosis of infection with human immunodeficiency virus (HIV).
* Pregnant women or nursing.
* Women of childbearing potential not using effective contraceptive method.
* Patients who are unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Every 8 weeks
  The primary endpoint is overall response rate, defined as the proportion of patients with response defined as complete or partial response according to RECIST CRITERIA 1.1 measured by an external evaluator

SECONDARY OUTCOMES:
Clinical benefit | Every 8 weeks
  Clinical benefit defined as stable disease for more than 6 months plus complete and partial response rates, measured by an external evaluator.
Progression-free survival | Every 8 weeks
  Progression-free survival is defined as the time since the start of treatment until progressive disease assessed (through evaluation by an external radiologist) according to RECIST 1.1, or death by any cause.
Overall survival | Untill death
  Overall survival, defined as the time since the start of treatment until the patient dies by any cause.
Quality of life | Every 4 weeks
  Quality of life measured by the validated in Spanish EORTC QLQ-C30 questionnaire.
Safety profile | Every 4 weeks
  Toxicities will be classified according to the NCI-CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Garcia-Donas, MD, Study Director — Hospital Universitario Fundación de Alcorcón, Servicio de Oncología Médica, c/ Budapest, 1,28922 Alcorcón (Madrid), Spain
Locations (10):
- Spain (10):
  - Complejo Hospitalario Universitario de Santiago de Compostela, Santiago de Compostela, A Coruña
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Reina Sofía, Córdoba, Cordoba
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital La Paz, Madrid, Madrid
  - Hospital Morales Meseguer, Murcia, Murcia
  - Complejo Hospitalario de Navarra, Navarra, Navarre
  - Hospital Son Llatzer, Palma de Mallorca, Palma de Mallorca
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario y Politécnico La Fe, Valencia, Valencia

REFERENCES:
- [Derived] Garcia-Donas J, Hurtado A, Garrigos L, Santaballa A, Redondo A, Vidal L, Lainez N, Guerra E, Rodriguez V, Cueva J, Bover I, Palacio I, Rubio MJ, Prieto M, Lopez-Guerrero JA, Rodriguez-Moreno JF, Garcia-Casado Z, Garcia-Martinez E, Taus A, de Castro IP, Navarro P, Grande E; Spanish Group for Research in Orphan, Infrequent Tumors (GETHI). Open-label phase II clinical trial of ketoconazole as CYP17 inhibitor in metastatic or advanced non-resectable granulosa cell ovarian tumors: the GREKO (GRanulosa Et KetOconazole) trial, GETHI 2011-03. Clin Transl Oncol. 2023 Jul;25(7):2090-2098. doi: 10.1007/s12094-023-03085-w. Epub 2023 Jan 28. PMID 36708371